CLINICAL TRIAL: NCT05953623
Title: A Phase Ib Dose-Escalation Study of Intra-arterial Albumin Infusion After Endovascular Therapy for Stroke Patients
Brief Title: Intra-arterial Albumin Infusion After Endovascular Therapy for Stroke Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tianjin Huanhu Hospital (Other)
Responsible Party: Principal Investigator, Ming Wei, Chief physician, Tianjin Huanhu Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJHH-2023-WeiMing617
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Stroke, Acute Ischemic; Albumin; Endovascular Procedures; Large Vessel Occlusion
Keywords: Acute Ischemic Stroke; Albumin; Endovascular Therapy; Large Vessel Occlusion
MeSH Terms: conditions — Ischemic Stroke | interventions — Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intra-arterial albumin infusion (Experimental)
  Interventions: Biological: Albumin

INTERVENTIONS:
Biological: Albumin — In the first phase of the study, a 3 + 3 dose-escalation study with 7 doses (0.25g/kg, 0.35g/kg, 0.40g/kg, 0.45g/kg, 0.5g/kg, 0.55g/kg, 0.60g/kg). Intra-arterial albumin infusion will be applied after successful recanalization of the culprit artery in the anterior circulation. In the second phase of the study, at the maximum safe dose determined in the first phase, an additional 15 to 20 patients will be enrolled for intra-arterial albumin infusion.

SUMMARY:
The purpose of this study is to investigate the safety and feasibility of intra-arterial albumin infusion for patients with acute ischemic stroke after successful thrombectomy and to further explore the optimal dose of albumin through the implementation of a 3 + 3 dose-escalation design. At the maximum safe dose determined in the 3+3 dose-escalation phase, an additional 15 to 20 patients will be enrolled in the study, and comparisons were made with external patients who received endovascular treatment alone.

DETAILED DESCRIPTION:
Albumin, the predominant plasma protein synthesized primarily in the liver, possesses various biochemical properties that are expected to confer a neuroprotective effect following acute ischemic stroke. Despite being utilized as a neuroprotective agent for stroke patients, albumin has not demonstrated efficacy, partly due to the persistence of the occluded vessel responsible for the stroke, thereby hindering the albumin's ability to exert its therapeutic effects in the ischemic region. In light of the advent of thrombectomy and subsequent recanalization of occluded blood vessels, it is imperative to reassess the potential impact of albumin. In first phase of this study, we plan to conduct a 3 + 3 dose-escalation trial to determine the safety and feasibility of intra-arterial albumin infusion for stroke patients undergoing successful mechanical thrombectomy. Since this is a 3 + 3 dose-escalation study with 7 doses (0.25g/kg, 0.35g/kg, 0.40g/kg, 0.45g/kg, 0.5g/kg, 0.55g/kg,0.60g/kg), a minimum of 21 (7 groups × 3 patient/group) patients will be required, assuming no major response occurs at any dose level, and a maximum of 42 (7 groups × 6 patient/group) patients will be required, assuming one major response occurs at each dose level. In second phase, at the maximum safe dose determined in the first phase, an additional 15 to 20 patients will be enrolled for intra-arterial albumin infusion.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years;
* Patients with acute ischemic stroke caused by large vessel occlusion in the intracranial anterior circulation (internal carotid artery, middle cerebral artery M1 and M2 segments) ;
* mTICI score ≥ 2b for the occlude vessel after mechanical thrombectomy;
* Baseline National Institutes of Health Stroke score (NIHSS) ≥ 6;
* Stroke onset to arterial puncture time within 24 hours.

Exclusion Criteria:

* Upon admission, the patient's medical history and physical examination revealed manifestations indicative of congestive heart failure (CHF), such as jugular venous distention, the presence of a third heart sound, resting tachycardia at a rate of 100 beats per minute attributable to heart failure, hepatomegaly, and/or lower extremity edema attributable to heart failure or of unknown etiology;
* History of acute myocardial infarction within the preceding 3 months;
* The patient's medical history, electrocardiogram findings upon admission, or physical examination indicated the presence of second- or third-degree heart block or any arrhythmia associated with hemodynamic instability, as determined by the investigator's assessment;
* Acute or chronic renal failure with serum creatinine levels exceeding 2.0 mg/dL;
* Severe anemia characterized by a hematocrit below 32%;
* Computed tomography findings upon admission indicating the presence of any form of hemorrhage;
* Pregnancy status;
* Previous history of allergic reactions to albumin administration;
* Elevated blood pressure exceeding 185/110 mmHg when investigating the use of albumin administration;
* Presence of other potentially life-threatening medical conditions;
* Individuals with current chronic lung diseases, such as chronic obstructive pulmonary disease, bronchiectasis, or any other lung disorder that significantly impairs daily activities; 12. Individuals with known allergies to albumin.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-06-29 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
All cause of death | 90 days after initiation of infusion of albumin intra-arterially.
  all cause of death within 90 days

SECONDARY OUTCOMES:
symptomatic intracranial hemorrhage | 24 (±6) hours after initiation of infusion of albumin intra-arterially
  symptomatic intracranial hemorrhage within 24 (±6) hours
rate of serious adverse events | 90 (±14) days after initiation of infusion of albumin intra-arterially
  rate of serious adverse events within 90 (±14) days
all intracranial hemorrhages | 24 (±6) hours after initiation of infusion of albumin intra-arterially
  all intracranial hemorrhages within 24 (±6) hours
pneumonia | 24 (±6) hours after initiation of infusion of albumin intra-arterially
  pneumonia within 24 hours after infusion
adverse events related to albumin infusion | 24 (±6) hours after initiation of infusion of albumin intra-arterially
  adverse events related to albumin infusion within 24 hours after infusion

OTHER OUTCOMES:
Imaging Biomarker | 24 (±6) hours after initiation of infusion of albumin intra-arterially
  image biomarker outcomes include Infarct volume at 24 (±6) hours
Imaging Biomarker | 24 (±6) hours after initiation of infusion of albumin intra-arterially
  Infarct volume growth from baseline at 24 (±6) hours
early neurological biomarkers | 24 (±6) hours after initiation of infusion of albumin intra-arterially;
  NIHSS scores at 24 (±6) hours
early neurological biomarkers | 7 (±1) days or at hospital discharge after initiation of infusion of albumin intra-arterially
  NIHSS scores at 7 (±1) days or at hospital discharge
long-term neurological biomarkers | 90 (±14) days after initiation of infusion of albumin intra-arterially
  Neurologic outcomes include proportion of mRS scores 0-2 at 90 (±14) hours
long-term neurological biomarkers | 90 (±14) days after initiation of infusion of albumin intra-arterially
  distribution of mRS scores at 90 (±14) days
peripheral immune responses | 24 (±6) hours after initiation of infusion of albumin intra-arterially.
  immune cell counts (neutrophil , white blood cell , lymphocyte , monocyte , platelet ) at 24 hours.
peripheral immune responses | 24 (±6) hours after initiation of infusion of albumin intra-arterially.
  inflammatory markers(neutrophil-to-lymphocyte ratio (NLR), platelet-to-lymphocyte ratio (PLR), and systemic immune-inflammation index (SII) )at 24 hours.
circulating molecular | 24 (±6) hours after initiation of infusion of albumin intra-arterially.
  Proteome and Metabolome analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Du K, Liu S, Nguyen TN, Pan S, Baron JC, Xu Y, Abdalkader M, Luo L, Wang S, Chen J, Dou Y, Liu S, Ji X, Wei M. Intra-arterial human serum albumin therapy following mechanical thrombectomy for acute ischemic stroke: the AMASS pilot trial. J Neurointerv Surg. 2025 Sep 8:jnis-2025-023998. doi: 10.1136/jnis-2025-023998. Online ahead of print. PMID 40921621
- [Derived] Pan S, Du K, Liu S, Wang S, Luo L, Xu Y, Cao C, Chen J, Ji X, Wei M. Albumin adjuvant therapy for acute ischemic stroke with large vessel occlusion (AMASS-LVO): rationale, design, and protocol for a phase 1, open-label, clinical trial. Front Neurol. 2024 Sep 30;15:1455388. doi: 10.3389/fneur.2024.1455388. eCollection 2024. PMID 39403266